CLINICAL TRIAL: NCT00004218
Title: Chronic Lymphocytic Leukemia Trial 4: A Randomized Comparison of Chlorambucil, Fludarabine and Fludarabine Plus Cyclophosphamide
Brief Title: Chemotherapy in Treating Patients With Newly Diagnosed Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Leukemia Research Fund (Other)
Collaborators: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067454; LRF-CLL4; LRG-MRC-LEUK-CLL4; EU-99030; MRC-LEUK-CLL4; EUDRACT-58585610; ISRCTN58585610; NCT00222599 (obsolete NCT alias)
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2006-01

CONDITIONS: Leukemia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Chlorambucil; Cyclophosphamide; Doxorubicin; fludarabine phosphate; Prednisolone; Vincristine

INTERVENTIONS:
Drug: chlorambucil
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: fludarabine phosphate
Drug: prednisolone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known which regimen of chemotherapy is more effective for chronic lymphocytic leukemia.

PURPOSE: This randomized phase III trial is studying chlorambucil to see how well it works compared to fludarabine and cyclophosphamide or fludarabine alone in treating patients with newly diagnosed chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival rate of patients with newly diagnosed chronic lymphocytic leukemia treated with chlorambucil alone vs fludarabine with or without cyclophosphamide.
* Compare the response rate and duration of remission in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Determine the impact of the drug response information provided by the DiSC assay on response rate and survival in relapsed or nonresponding patients.
* Assess the prognostic value of five genetic markers: trisomy 12 and deletions at 11q23, 13q14, p53, and 6q21 in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients enter one of three treatment arms in the first randomization. Depending on response, some patients may also participate in a second randomization to one of two treatment arms.

* First randomization:

  * Arm I: Patients receive oral chlorambucil daily for 7 days. Treatment repeats every 4 weeks until maximum response or up to 1 year.
  * Arm II: Patients receive fludarabine IV or orally daily for 5 days. Treatment repeats every 4 weeks for 3-8 courses.
  * Arm III: Patients receive cyclophosphamide IV and fludarabine IV for 3 days or orally daily for 5 days. Treatment repeats every 4 weeks for 3-8 courses.

Patients who relapse after being in remission for at least 1 year may repeat the initial therapy or may participate in a second randomization. Patients who experience progressive disease or relapse within 1 year after treatment proceed to a second randomization.

* Second randomization:

  * Arm I: Treatment is guided by the results of the DiSC assay. Treatment may be one of the first-line treatments with fludarabine or standard CHOP chemotherapy repeated every 4 weeks (cyclophosphamide IV, doxorubicin IV, vincristine IV, and oral prednisolone on days 1-5) or any other therapy guided by the results of the DiSC assay.
  * Arm II: Treatment is physician's choice, which may include any of the options in arm I.

Quality of life is assessed prior to initial therapy; at 3, 6, and 12 months; and then annually thereafter.

Patients are followed annually for survival.

PROJECTED ACCRUAL: A total of 750 patients will be accrued for this study within 6-7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia (CLL) requiring therapy and meeting the following criteria:

  * Previously untreated disease
  * Peripheral blood morphology, excluding other leukemia and low-grade lymphoma in leukemic phase
  * Cell markers: CD5+, CD23+, SmIg (weak), CD79b-, FMC7-
  * Persistent lymphocytosis (greater than 10,000/mm^3)
  * At least 40% bone marrow infiltration
* Stage 0 or I progressive disease indicated by at least one of the following:

  * Persistent rise in lymphocyte count with doubling time less than 12 months
  * Downward trend in hemoglobin and/or platelet count
  * At least 50% increase in size of liver and/or spleen and/or lymph nodes
  * Appearance of lymphadenopathy, hepatomegaly, or splenomegaly
  * Constitutional symptoms caused by disease

    * Pyrexia
    * Night sweats
    * Weight loss OR
* Stage II or III

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)*
* SGOT/SGPT no greater than 2 times ULN* NOTE: * Unless due to CLL

Renal:

* Creatinine clearance at least 30 mL/min

Other:

* No other cancer or life-threatening disease
* Not pregnant
* Fertile patients must use effective contraception during and for 6 months after study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No concurrent corticosteroids (e.g., dexamethasone) as antiemetics

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Catovsky, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (86):
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Alvarez, Buenos Aires
- University Hospital Rebro, Zagreb, Croatia
- Greece (2):
  - University of Ioannina, Ioannina
  - University of Patras Medical School, Rio Patras
- Ireland (2):
  - St. James' Hospital, Dublin
  - Galway University Hospital, Galway
- Ospedali Riuniti di Bergamo, Bergamo, Italy
- Canterbury Health Laboratories, Christchurch, New Zealand
- Russian Academy of Medical Sciences Cancer Research Center, Moscow, Russia
- United Kingdom (76):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - Horton Hospital, Banbury, England
  - North Hampshire Hospital, Basingstoke, England
  - Selly Oak Hospital at University Hospital NHS Trust, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bradford Hospitals NHS Trust, Bradford, England
  - Royal Sussex County Hospital, Brighton, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - St Helier Hospital, Carshalton, England
  - Countess of Chester Hospital, Chester, England
  - Chesterfield Royal Hospital, Chesterfield, England
  - Saint Richards Hospital, Chichester, England
  - Darlington Memorial, Darlington, England
  - Dartford & Gravesham NHS Trust, Joyce Green Hospital, Dartford Kent, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Russells Hall Hospital, Dudley, England
  - Bishop Auckland Hospital, Durham, England
  - Epsom General Hospital, Epsom Surrey, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Queen Elizabeth Hospital, Gateshead-Tyne and Wear, England
  - Gloucester Royal NHS Trust - Glouchester Royal Hospital, Gloucester, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Harrogate District Hospital, Harrogate, England
  - Hemel Hempstead General, Hemel Hempstead, England
  - Institute of Oncology and Radiology of Serbia, High Wycombe, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Hull Royal Infirmary, Hull, England
  - Clinical Trials and Research Unit of the University of Leeds, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool and Broadgreen Hospitals, Liverpool, England
  - Walton General Hospital, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Whipps Cross Hospital, London, England
  - Royal Free and University College Medical School, London, England
  - Guy's and St. Thomas' Hospitals NHS Foundation Trust, London, England
  - St. George's Hospital, London, England
  - Royal Marsden NHS Foundation Trust - London, London, England
  - West Middlesex Hospital, Middlesex, England
  - Northern Cancer Network, Newcastle upon Tyne, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Bassetlaw Hospital & Community Services NHS Trust, Nottinghamshire, England
  - Farnborough Hospital, Orpington Kent, England
  - Wharfdale General Hospital, Otley, England
  - Pontefract General Infirmary, Pontefract West Yorkshire, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Oldchurch Hospital, Romford, England
  - Rotherham District General Hospital - NHS Trust, Rotherham, England
  - Conquest Hospital, Saint Leonards-on-Sea, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Royal South Hants Hospital, Southampton, England
  - Southampton General Hospital, Southampton, England
  - Staffordshire General Hospital, Stafford, England
  - North Staffs Royal Infirmary, Stoke-on-Trent, England
  - St. Peter's Hospital NHS Trust, Surrey, England
  - Torbay Hospital, Torquay Devon, England
  - City Hospital - Birmingham, West Bromwich, England
  - Good Hope Hospital Trust, West Midlands, England
  - Worthing Hospital, Worthing, England
  - Cancer Care Centre at York Hospital, York, England
  - Belfast City Hospital Trust, Belfast, Northern Ireland
  - Ulster Hospital, Dundonald, Northern Ireland
  - Craigavon Area Hospital, Portadown, Craigavon, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Monklands General Hospital, Airdrie, Scotland
  - Dumfries Royal Infirmary, Dumfries, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Southern General Hospital, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Victoria Hospital, Kirkcaldy, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Nevill Hall Hospital, Gwent, Wales
  - Singleton Hospital, Swansea, Wales

REFERENCES:
- [Result] Else M, Cocks K, Crofts S, Wade R, Richards SM, Catovsky D, Smith AG; UK National Cancer Research Institute (NCRI) Chronic Lymphocytic Leukaemia Trials Group. Quality of life in chronic lymphocytic leukemia: 5-year results from the multicenter randomized LRF CLL4 trial. Leuk Lymphoma. 2012 Jul;53(7):1289-98. doi: 10.3109/10428194.2011.649479. Epub 2012 Mar 1. PMID 22168274
- [Result] Gonzalez D, Martinez P, Wade R, Hockley S, Oscier D, Matutes E, Dearden CE, Richards SM, Catovsky D, Morgan GJ. Mutational status of the TP53 gene as a predictor of response and survival in patients with chronic lymphocytic leukemia: results from the LRF CLL4 trial. J Clin Oncol. 2011 Jun 1;29(16):2223-9. doi: 10.1200/JCO.2010.32.0838. Epub 2011 Apr 11. PMID 21483000
- [Result] Wade R, Di Bernardo MC, Richards S, Rossi D, Crowther-Swanepoel D, Gaidano G, Oscier DG, Catovsky D, Houlston RS. Association between single nucleotide polymorphism-genotype and outcome of patients with chronic lymphocytic leukemia in a randomized chemotherapy trial. Haematologica. 2011 Oct;96(10):1496-503. doi: 10.3324/haematol.2011.043471. Epub 2011 Jun 9. PMID 21659360
- [Result] Oscier D, Wade R, Davis Z, Morilla A, Best G, Richards S, Else M, Matutes E, Catovsky D; Chronic Lymphocytic Leukaemia Working Group, UK National Cancer Research Institute. Prognostic factors identified three risk groups in the LRF CLL4 trial, independent of treatment allocation. Haematologica. 2010 Oct;95(10):1705-12. doi: 10.3324/haematol.2010.025338. Epub 2010 May 29. PMID 20511662
- [Result] Else M, Smith AG, Cocks K, Richards SM, Crofts S, Wade R, Catovsky D. Patients' experience of chronic lymphocytic leukaemia: baseline health-related quality of life results from the LRF CLL4 trial. Br J Haematol. 2008 Dec;143(5):690-7. doi: 10.1111/j.1365-2141.2008.07407.x. Epub 2008 Oct 18. PMID 19016733
- [Result] Catovsky D, Richards S, Matutes E, Oscier D, Dyer M, Bezares RF, Pettitt AR, Hamblin T, Milligan DW, Child JA, Hamilton MS, Dearden CE, Smith AG, Bosanquet AG, Davis Z, Brito-Babapulle V, Else M, Wade R, Hillmen P; UK National Cancer Research Institute (NCRI) Haematological Oncology Clinical Studies Group; NCRI Chronic Lymphocytic Leukaemia Working Group. Assessment of fludarabine plus cyclophosphamide for patients with chronic lymphocytic leukaemia (the LRF CLL4 Trial): a randomised controlled trial. Lancet. 2007 Jul 21;370(9583):230-239. doi: 10.1016/S0140-6736(07)61125-8. PMID 17658394
- [Result] Dearden CE, Wade RL, Else M, et al.: The combination of fludarabine and cyclophosphamide has a beneficial effect on the incidence of hemolytic anemia in chronic lymphocytic leukemia: results from the UK LRF CLL4 trial. [Abstract] Blood 110 (11): A-2044, 2007.
- [Derived] Skowronska A, Parker A, Ahmed G, Oldreive C, Davis Z, Richards S, Dyer M, Matutes E, Gonzalez D, Taylor AM, Moss P, Thomas P, Oscier D, Stankovic T. Biallelic ATM inactivation significantly reduces survival in patients treated on the United Kingdom Leukemia Research Fund Chronic Lymphocytic Leukemia 4 trial. J Clin Oncol. 2012 Dec 20;30(36):4524-32. doi: 10.1200/JCO.2011.41.0852. Epub 2012 Oct 22. PMID 23091097